CLINICAL TRIAL: NCT04336085
Title: Comparison of Ultrasound Guided Caudal Block and Ultrasound Guided Pericapsular Nerve Group Block for Pediatric Hip Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: pericapsular nerve group block
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Post Operative Pain After Pediatric Hip Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- caudal group (Experimental): Caudal block using ultrasound guidance. the sacral hiatus will be visualized at the level of the sacral cornus by employing the linear transducer of ultrasound machine and the depth and gain will be adjusted for optimal visual quality.the needle will be advanced toward the upper third of the sacrococcygeal ligament. The needle advancement will be terminated immediately after penetrating the sacrococcygeal ligament.
  Interventions: Procedure: caudal block
- PENG group (Experimental): The ilio-pubic eminence (IPE), the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle will be visualized using a linear ultrasound probe. the needle will be introduced in a lateral to medial fashion in an in-plane approach to place the tip of the needle in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly.
  Interventions: Procedure: pericapsular nerve group block

INTERVENTIONS:
Procedure: caudal block — Caudal block will be performed using ultrasound guidance, the sacral hiatus will be visualized at the level of the sacral cornus by employing the linear transducer of ultrasound machine the ultrasound transducer will be rotated to 90 degree to obtain longitudinal views of the sacrococcygeal ligament and sacral hiatus and will be subsequently placed between the two cornua. The needle advancement will be terminated immediately after penetrating the sacrococcygeal ligament.
  Arms: caudal group
Procedure: pericapsular nerve group block — In PENG group, the patient will be placed in supine position. The ilio-pubic eminence (IPE), the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle will be visualized using a linear ultrasound probe. A 22-gauge, 50-mm needle will be introduced in a lateral to medial fashion in an in-plane approach to place the tip of the needle in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. Following negative aspiration, a total volume of 0.5 mL/kg local anesthetic solution will be injected.
  Arms: PENG group

SUMMARY:
Surgical repair of the hip can be extremely painful and is associated with considerable postoperative pain in children despite the use of systemic opioids. These patients may benefit from neuraxial analgesia in adjunction with general anesthesia. The reported advantages of this technique include decreased opiate exposure, decreased time in the post-anesthesia recovery room, decreased hospital stay, reduce the post-operative morbidity, provide early mobilization. Ultrasound guided caudal block has many advantages as it is helpful for visualization of the sacral hiatus, sacrococcygeal ligament, epidural space and the distribution of the local anesthetic agent within the epidural space. So, the success rate of caudal block is increase .

Pericapsular nerve group (PENG) block has been recently recommended by Girón-Arango et al. for use as postoperative analgesia in hip surgeries (8) It is a new regional anesthesia method in the region between the anterior inferior iliac spine (AIIS) and ilio-pubic eminence

DETAILED DESCRIPTION:
Surgical repair of the hip can be extremely painful and is associated with considerable postoperative pain in children despite the use of systemic opioids. These patients may benefit from neuraxial analgesia in adjunction with general anesthesia. The reported advantages of this technique include decreased opiate exposure, decreased time in the post-anesthesia recovery room, decreased hospital stay, reduce the post-operative morbidity, provide early mobilization. (1,2) Single shot caudal block has been the widely used to provide intraoperative and postoperative analgesia especially in pediatric surgery below the umbilical level, by block the region between T10 and S5 dermatomes. (3,4) The success rate of classic caudal epidural anesthesia method in pediatric patients has been reported to be about 75%. (5) Because there are many anatomical variations have been reported for sacral hiatus and sacral cornua.

Ultrasound guided caudal block has many advantages as it is helpful for visualization of the sacral hiatus, sacrococcygeal ligament, epidural space and the distribution of the local anesthetic agent within the epidural space. So, the success rate of caudal block is increase (6) However caudal block has adverse effects such as hypotension, postoperative nausea, vomiting, urinary retention, excessive motor block, and pruritus that limit the use of caudal block in children. (7) Regional anesthetic techniques seem to be a better choice for improving acute pain management in these patients, with fewer adverse effects. Pericapsular nerve group (PENG) block has been recently recommended by Girón-Arango et al. for use as postoperative analgesia in hip surgeries (8) It is a new regional anesthesia method in the region between the anterior inferior iliac spine (AIIS) and ilio-pubic eminence (IPE).

The anterior capsule is the most richly innervated section of the joint suggesting these nerves should be the main targets for hip analgesia. (9) To the best of our knowledge, there are no previously published data comparing the pericapsular nerve group (PENG) block with caudal block techniques.

ELIGIBILITY:
Inclusion Criteria:

* 1- American Society of Anaestheologists physical activity class I and II. 2-aged between 1 year to 6 years. 3- undergoing pediatric elective hip surgery.

Exclusion Criteria:

* 1-Children with severe systemic disease with American Society of Anaestheologists physical activity class III or IV.

  2-children with previous neurological or spinal disorders. 3-coagulation disorder. 4-infection at the block injection site. 5-history of allergy to local anesthetics. 6-bilateral hip surgery.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Total doses of postoperative analgesic requirement | postoperative first day
  Total doses of postoperative morphine analgesic requirement

SECONDARY OUTCOMES:
Evaluation of the pain scores | postoperative first day
  Evaluation of the pain scores by FLACC scale
Time to first rescue analgesic demand after surgery | postoperative first day

CONTACTS AND LOCATIONS:
Locations (1):
- Tarek Abdel Hay, Tanta, El Gharbyia, Egypt

IPD SHARING:
Plan to Share IPD: No